CLINICAL TRIAL: NCT06193798
Title: Diagnostic Laparoscopy For Unexplained Abdominal Pain Risks &Benefits
Brief Title: Diagnostic Laparoscopy for Unexplained Abdominal Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nouran, Nouran Mohsen abdelshakour, Assiut University
Other Study IDs: Diagnostic laparoscopy
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-12

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evalute the efficiency and safety of diagnostic laparoscopy for patients who have unexplained abdominal pain after completing all needed imaging and laboratories in general surgery depatment Assuit university hospital

DETAILED DESCRIPTION:
Abdominal pain may be a simple thing or it may be a dangerous and life threatening one.It is very difficult to come to a correct diagnosis(1).Diagnostic laparoscopy gives many advantages in the management of many intra-abdominal conditions where the correct diagnosis could not establish clinically or even with the help of imaging studies(2).Diagnostic laparoscopy can be done under direct vision using simple instruments of laparoscopy. With advances in optics, laparoscopy allows visualization of entire peritoneal cavity and further makes possible histological diagnosis of target biopsy under vision(3).In case of diagnostic uncertainty, laparoscopy may help to avoid unnecessary laparotomy, provides accurate diagnosis, helps to plan surgical treatment, improves the outcome in the majority of patients with abdominal pain and allows surgeons to diagnose and treat many abdominal conditions that cannot be properly managed otherwise(4).Many factors like high diagnostic yield, its applicability and therapeutic management in both elective and emergency setups, reduced hospital stay, low morbidity, and expenditure have made this treatment modality most popular(5). On the otherhand there are Complications related to laparoscopic surgery up to one-half of complications occur at the time of abdominal access for camera or port placement , Others arise from abdominal insufflation, tissue dissection, and hemostasis .Conversion to an open procedure may be needed to manage complications (6).Recent treatises deficient in evalution of the role of lap in cases with vague abdominal pain for this the interest of our study is to evalute the efficiency and safety of diagnostic laparoscopy for patients who have unexplained abdominal pain after completing all needed imaging and laboratories.

ELIGIBILITY:
Inclusion Criteria:

* Patients with obscure abdominal pain
* Age from 18 years old up to 70 years old

Exclusion Criteria:

1. Current use of narcotics
2. patients have uncontrolled coagulopathy
3. Patients are Haemodynamically unstable
4. patients have Cardiopulmonary problems
5. Patients refusing the diagnostic laparoscopy after routine investigations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To evalute the efficiency and safety of diagnostic laparoscopy for unexplained abdominal pain cases in general surgery depatment Assuit university hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic laparoscopy for unexplained abdominal pain | Diagnostic laparoscopy
  For diagnosis any obscure abdominal pain

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Hamed, Study Director — Assiut University

REFERENCES:
- [Background] Ning N, Xia SY, Ma B, Li R, DU XH. [Application of laparoscopic technique in acute abdomen of gastrointestinal surgery]. Zhonghua Wei Chang Wai Ke Za Zhi. 2013 Oct;16(10):960-2. Chinese. PMID 24158868